CLINICAL TRIAL: NCT02819505
Title: The Effects of 4 Week β-alanine Supplementation on Knee Extensor Contractile and Force Properties in Active Male Adults (18-30 Years).
Brief Title: β-alanine Supplementation on Knee Extensor Contractile and Force Properties
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, Rebecca Louise Stannard, Academic Associate, Nottingham Trent University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 369
Record Dates: First submitted 2016-06-21; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Muscle Function
Keywords: beta-alanine; carnosine; neuromuscular; stimulation; skeletal muscle
MeSH Terms: interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beta-alanine supplementation (Experimental): Participants will be supplemented with 6.4g·d-1 β-alanine (CarnoSyn™, NAI, USA). The β-alanine dosing regimen will consist of two 800 mg tablets four times per day at 3-4 hour intervals or the same regimen for placebo tablets. The use of multiple small doses throughout the day has been used in numerous studies using β-alanine in solutions or gelatine capsules (Hoffman et al., 2008; Sale et al., 2011; Saunders et al., 2012; Sale et al., 2012; Tobias et al., 2013) in order to circumvent potential symptoms of paraesthesia (see box xii for possible risks and discomforts). Overall increases have been shown to be between 40% and 80% depending upon dose (between 3.2 and 6.4 g·d-1) and duration of administration (between 4 and 10 weeks) (Sale et al., 2012).
  Interventions: Dietary Supplement: beta-alanine
- Placebo supplementation (Placebo Comparator): Participants will be supplemented with 6.4g·d-1 placebo (maltodextrin; NAI, USA).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: beta-alanine
  Arms: Beta-alanine supplementation
Dietary Supplement: Placebo
  Arms: Placebo supplementation

SUMMARY:
Carnosine (made by bonding β-alanine and histidine) has been suggested to contribute to the extension of physical exercise, counteracting the decline in muscle performance due to fatigue. However this process is largely restricted by the levels of β-alanine available in the human body. Carnosine levels can be raised through long term ingestion of food products, such as meat, fish and poultry, however it can also be significantly increased by β-alanine supplementation. Improved β-alanine levels can potentially advance exercise capacity and exercise performance, which may have been previously limited. Recently research has demonstrated no beneficial effect of β-alanine supplementation on neuromuscular performance in active, healthy males when they were well rested, with no prior exercise or fatigue of the assessed muscle. It remains unknown if β-alanine supplementation would aid physical performance when the muscle has already been fatigued. This is currently being investigated in older adults (60-80 years), however there is no clear comparison between the potential effects in younger and older participants.

Therefore this investigation hopes to examine the effects of 4 week β-alanine supplementation on lower limb contractile and force properties, pre and post muscle specific fatigue in 18-30 year old males.

DETAILED DESCRIPTION:
Carnosine (β-alanyl-L-histidine) is a naturally occurring dipeptide formed by bonding histidine and β-alanine in a reaction catalysed by carnosine synthase. One role of carnosine within the human system, is as an intracellular pH buffer due to its pKa of 6.83. Carnosine is suitable over the whole exercise induced intramuscular pH transit-range. Carnosine in untrained populations can neutralise 2.4 to 10.1mmol H+.kg-1 of dry mass muscle as intramuscular pH declines, adding at least 7% to 10% to total intramuscular buffering capacity. It has also been argued that carnosine in combination with anserine can contribute as much as 40% to the buffering capacity between pH ranges of 6.5 to 7.5. β-alanine has been suggested as the rate limiting factor for muscle carnosine synthesis, through ingestion of β-alanine in diet (meat, fish and poultry) or via short-term supplementation, demonstrating significant increases in muscle carnosine concentrations. Increases in carnosine concentrations between 40% and 80% have been shown, depending upon dose (between 3.2 and 6.4 g·d-1) and duration of administration (between 4 and 10 weeks). Increasing β-alanine concentrations therefore enhance carnosine synthesis with the muscle fibers and improves intramuscular buffering capacity. Exercise performance and capacity measurements that previously were limited by the accumulation of H+ have been demonstrated significant improvements through supplementation with β-alanine.

Research already conducted at Nottingham Trent University and approved by this ethical advisory committee has demonstrated no significant effect of β-alanine supplementation on neuromuscular performance in healthy, active males. However, this research was conducted with well rested participants, with no prior exercise or fatigue of the assessed muscle; therefore there was no accumulation of H+ demonstrated within the muscle. These previous investigations are therefore contemplating how β-alanine supplementation alters performance when intramuscular buffering has not been altered (at the start of the exercise), whereas the proposed study will examine the effect of β-alanine supplementation on performance when intramuscular pH has already been challenged (due to fatiguing exercise). It is hypothesised that β-alanine supplementation over 4 weeks will beneficially alter the contractile and force properties of the muscle fibres within the lower limb muscles, improving physical performance when the muscle is already fatigued.

Aims of the project:

To examine the effects of 4 week β-alanine supplementation on knee extensor contractile and force properties, pre and post induced muscle specific fatigue in 18-30 year old males.

ELIGIBILITY:
Inclusion Criteria:

* physically active
* male

Exclusion Criteria:

* vegetarian/vegan
* have been using β-alanine or carnosine supplements within the past 6 months
* Bone disorders in the assessed lower limb, sustained within the previous 2 years, including osteoarthritis, osteoporosis, bone cyst and osteopenia.
* Non-arthroscopic joint surgery, or joint replacement, ever, in the assessed limb (knee, hip and ankle).
* Lower limb leg injuries including sprains and strains, joint dislocations and fractures.
* Regular knee pain in the assessed limb when performing daily movement tasks.
* Participation within a resistance training programme in the last 6 months

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Half relaxation time | 4 weeks
  The time taken to decline to 50% maximum following a evoked twitch contraction

SECONDARY OUTCOMES:
Force frequency relationship | 4 weeks
  Assessed during electrically evoked contractions.
Time to peak tension | 4 weeks
  The time taken to reach peak in evoked twitch contractions
Electromechanical delay | 4 weeks
  The time between EMG onset and force onset in twitch contractions
Maximal voluntary force production | 4 weeks
  The maximal force produced during a voluntary isometric contraction
Explosive voluntary force production | 4 weeks
  The quickest rate of force developed during voluntary isometric contractions at greater than 80% of voluntary maximum, with no pre-tension or swinging back of the assessed leg.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sale C, Saunders B, Harris RC. Effect of beta-alanine supplementation on muscle carnosine concentrations and exercise performance. Amino Acids. 2010 Jul;39(2):321-33. doi: 10.1007/s00726-009-0443-4. Epub 2009 Dec 20. PMID 20091069
- [Background] Sale C, Artioli GG, Gualano B, Saunders B, Hobson RM, Harris RC. Carnosine: from exercise performance to health. Amino Acids. 2013 Jun;44(6):1477-91. doi: 10.1007/s00726-013-1476-2. Epub 2013 Mar 12. PMID 23479117
- [Background] Harris RC, Sale C. Beta-alanine supplementation in high-intensity exercise. Med Sport Sci. 2012;59:1-17. doi: 10.1159/000342372. Epub 2012 Oct 15. PMID 23075550
- [Background] Artioli GG, Gualano B, Smith A, Stout J, Lancha AH Jr. Role of beta-alanine supplementation on muscle carnosine and exercise performance. Med Sci Sports Exerc. 2010 Jun;42(6):1162-73. doi: 10.1249/MSS.0b013e3181c74e38. PMID 20479615
- [Derived] Jones RL, Barnett CT, Davidson J, Maritza B, Fraser WD, Harris R, Sale C. beta-alanine supplementation improves in-vivo fresh and fatigued skeletal muscle relaxation speed. Eur J Appl Physiol. 2017 May;117(5):867-879. doi: 10.1007/s00421-017-3569-1. Epub 2017 Mar 27. PMID 28349262